CLINICAL TRIAL: NCT05687175
Title: Study to Translate and Determine the Validity and Reliability of Malay Version of painDETECT Questionnaire (PDQ-M)
Brief Title: Translation and Validation of Malay Version of painDETECT Questionnaire
Acronym: PDQM
Status: Completed | Type: Observational
Sponsor: University Malaysia Sarawak (Other)
Collaborators: Persatuan Diabetes Malaysia (Unknown)
Responsible Party: Sponsor
Other Study IDs: PDQ-M
Record Dates: First submitted 2023-01-06; First posted 2023-01-18 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Neuropathic Pain, Nociceptive Pain
MeSH Terms: conditions — Neuralgia; Nociceptive Pain | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neuropathic pain: Questionnaire administration and socio-demographic data collection
  Interventions: Other: Questionnaire
- Nociceptive pain: Questionnaire administration and socio-demographic data collection
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — Questionnaire administration (PDQ-M, NRS, SF-36)

SUMMARY:
The translation and cultural adaptation process of the English version of PDQ will be performed based on international guidelines. Subsequently, patients with neuropathic and nociceptive pain based on clinician's diagnoses will be recruited to complete three-type numeric rating scale (NRS) of pain followed by PDQ-M and SF-36 questionnaire. Patients' socio-demographic data and clinical characteristics will be reported using frequency for categorical variables and mean with standard deviation for continuous variables. Normality will be assessed using Shapiro Wilk test and histograms for continuous variables. Data will be compared between groups using chi-square test (for categorical variables) and t-test or Mann-Whitney's U test (for continuous variables). Suitability of PDQ-M data for factor analysis will be verified using the Bartlett's test of sphericity and the Kaiser-Mayer-Olkin (KMO) measure of sampling adequacy. Parallel analysis will performed to obtain the suitable factors. Construct validity will be investigated by exploratory factorial analysis (EFA) with varimax rotation. A factor loading of >0.40 will be used to determine the items for each factor. The internal consistency of the questionnaire will be assessed using Cronbach's alpha test. A p value of <0.05 is taken as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* able to read and understand the Malay language
* diagnosed to have neuropathic or nociceptive pain by clinician
* stable disease condition
* pain duration of at least 4 weeks

Exclusion Criteria:

* acute illness
* poor mental health status that prevents them from understanding or responding to the proposed questions
* cultural or language barrier

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have been diagnosed to have neuropathic or nociceptive pain by clinicians, with stable disease condition and pain duration of at least 4 weeks prior to recruitment.
Sampling Method: Probability Sample
Enrollment: 97 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
PDQ-M scores | 2-5 weeks
  Total of PDQ-M scores

CONTACTS AND LOCATIONS:
Locations (4):
- Malaysia (4):
  - Penang General Hospital, Pulau Pinang, Pulau Pinang
  - Sarawak General Hospital, Kuching
  - Malacca General Hospital, Malacca
  - Putrajaya Hospital, Putrajaya